CLINICAL TRIAL: NCT01644708
Title: Th Efficacy of Individual Empowerment on Overweight and Obese Patients - a Prospective Observational Study.
Brief Title: Empowerment and Overweight - a Prospective Observational Study
Acronym: ADPB-EMPW
Status: Completed | Type: Observational
Sponsor: Azienda Per I Servizi Sanitari N. 2 Isontina (Other)
Collaborators: Azienda per i servizi Sanitari 4 Medio Friuli, Dipartimento di Salute Mentale, Udine (Unknown); Associazione Diamo Peso al Benessere (Unknown); Università degli Studi di Udine, Facoltà di Medicina e Chirurgia, Clinica Psichiatrica (Unknown); Centro Regionale di Formazione per l'Area delle Cure Primarie (Unknown)
Responsible Party: Principal Investigator, Pierluigi Struzzo, MD, Research Area Responsible, Azienda Per I Servizi Sanitari N. 2 Isontina
Other Study IDs: CeformedDSM1
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Overweight; Obesity; Power, Personal
Keywords: Obesity; Overweight; Individual empowerment; Physical parameters; Self esteem
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Overweight, obese adult patients: Patients following a self empowerment group will be included in the study
  Interventions: Behavioral: Self empowerment

INTERVENTIONS:
Behavioral: Self empowerment — 1. Group meeting, introducing the method and the assessment tools
  1. Self-empowerment,
  2. Handing over the "journal",
  3. Questionnaire about emotional states and motivations for losing weight and for change.
  The group meetings, lasting one hour and a half, will take place every week, always on the same day and at the same time, for one year. During each meeting the participant "weighs himself" and he notes his weight down in his journal.
  Other Names: self-empowerment; self-esteem

SUMMARY:
Overweight and obesity put an heavy burden over people's health. Many methods are reported in medical literature but none of them proved to be effective in maintaining the results achieved over time. Motivational change remains a fundamental step towards the maintenance of a new lifestyle. Strengthening personal capabilities and self-esteem seem to be key strategies in motivating persons for change and facilitating a capacity of coping.

The aim of this study is to observe the effects of an individual empowerment program on the health of a group of overweight/obese persons.

DETAILED DESCRIPTION:
With this observational, uncontrolled prospective study we aim to observe any clinical modifications (concerning weight and other health indicators) achieved by a group of overweight and obese persons who underwent a therapy treatment by means of "self-empowerment".

The study will include all adults, with a Body Mass Index (BMI) above 25, entering the new "therapy groups" of the project, named "Diamo Peso al Benessere" ("Let's Give Weight to Well-Being") an NGO located within the Local Health Unit 4 Medio Friuli, Mental Health Department.

The added value of the strategy proposed by this association is relevant because it is mainly directed to the the improvement of the capacity building of each obese participant instead of focusing only to the food intake. General practice trainees will be dedicated to the evaluation and monitoring of the health status of a group of obese patients included into self-empowerment groups will be assessed for the following year. Major health indicators will be assessed: Body weight, height, waist circumference, brachial blood pressure (two measurements), non-invasive oxymetry.

Some questionnaires will be utilized: Antonovsky's sense of coherence scale, 10-point Likert scale about empowerment, Likert scale about perceived health, Berlin test, Hamilton rating scale for depression.

Blood tests will also be observed. Statistical Analysis A descriptive analysis of all the parameters collected, both the baseline data and those from the 6 and 12- month follow-ups.

For continuous variables (age, weight, BMI…) indicators will be calculated such as the mean, standard deviation, minimum, median and maximum values. The categorical data will be presented by means of frequency tables (n, %).

The changes in the parameters and in the distribution of categorical variables pertaining to the main and secondary outcomes will be assessed by comparing the baseline data collected and those from the 6 and 12-month follow-ups. McNemar's test will be used on the categorical variables, with a level of significance for the p-value fixed at < 0.05. This will allow to record any differences in the distributions of the main factors of interest. T-tests will be used for paired data for assessing changes in the categorical variables.

ELIGIBILITY:
Inclusion Criteria:

- The study will include all adults, with a Body Mass Index (BMI) above 25, entering the new "therapy groups" of the project, named "Diamo Peso al Benessere" ("Let's Give Weight to Well-Being"), (Local Health Unit 4 Medio Friuli, Mental Health Department). Before being included in the therapy groups, persons will undergo three individual in-depth interviews with an empowerment consultant, with:

* Verification of the motivation (Importance of the problem + Self-esteem, Likert scales 0 -10)
* Request to underwrite the "therapy contract"
* Final meeting for inclusion in the group and acquisition of informed consent.

Exclusion Criteria:

- minors will be excluded and

* those who must shed weight in a short time because of planned surgery,
* those who suffer from severe health problems (severe stroke outcomes, heart or kidney failure, neoplasia)
* those who want to lose weight only for esthetic reasons,
* those who cannot guarantee regular weekly attendance for the treatment,
* those who also use other means for losing weight (weight-loss surgery, psychoanalysis, or other nutritional regimens).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult persons with BMI equal or above 25
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Decreasing body weight | 6,12 months
  A persistent reduction of body weight is expected after 6 and 12 months

SECONDARY OUTCOMES:
Improved blood pressure control | 6 and 12 months
decreasing glycemic levels | 6 and 12 months
decreasing total cholesterol values | 6 and 12 months
decreasing triglyceride values | 6 and 12 months
improvements in the creatinine levels | 6 and 12 months
stabilization and improvement of mood and temper (reduction in benzodiazepines and antidepressants) | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Struzzo, MD, Principal Investigator — Regional Centre for the Training in Primary Care; Mario Novello, MD, Study Director — Azienda per i Servizi Sanitari Medio Friuli; Anita Cacitti, dr, Study Chair — Azienda per i Servizi Sanitari Medio Friuli
Locations (1):
- Dipartimento di Salute Mentale, Udine, Italy

REFERENCES:
- [Derived] Struzzo P, Fumato R, Tillati S, Cacitti A, Gangi F, Stefani A, Torcutti A, Crapesi L, Tubaro G, Balestrieri M. Individual empowerment in overweight and obese patients: a study protocol. BMJ Open. 2013 May 14;3(5):e002669. doi: 10.1136/bmjopen-2013-002669. PMID 23676799